CLINICAL TRIAL: NCT03188601
Title: Relative Inactivity of Alpha-1-antitrypsin After Bone Marrow Transplantation as a Dynamic Biomarker for GVHD and Prognosis: a Prospective Cohort Study
Brief Title: α1-antitrypsin (AAT) Levels and Functions in Allogeneic Bone Marrow Transplantation and Throughout Progression Into GVHD
Acronym: AATGVHD-MARK
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Soroka University Medical Center (Other); Tel-Aviv Sourasky Medical Center (Other Government); Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0196-17-RMB; A1373 (Other Grant/Funding Number: Rosetrees trust)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: GVHD; Bone Marrow Transplant Failure; Alpha 1-Antitrypsin
Keywords: Graft vs Host Disease; Immune System Diseases; Protease Inhibitors; Alpha 1-Antitrypsin; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Trypsin Inhibitors; Serine Proteinase Inhibitors
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Graft vs Host Disease; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum samples and peripheral blood mononuclear cells' RNA extracts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Rambam: Approximately 40 patients in total.No intervention planned.
- Soroka: Approximately 10 patients in total.No intervention planned.
- Tel Aviv Souraski: Approximately 40 patients in total.No intervention planned.
- Jerusalem Hadassah: Approximately 50 patients in total. No intervention planned.

SUMMARY:
Create a personalized time and context curve of patient circulating α1-antitrypsin (AAT) levels and functions before hematopoietic stem cell transplantation and throughout progression into GVHD.

PRIMARY ENDPOINT 1. Serum AAT levels and activity, before myeloablative preconditioning, as well as on days (-3),0,7,14,28 from HSCT and every 21 days thereafter.

SECONDARY ENDPOINTS 1. Correlation between AAT patterns and:

* Circulating immune cell activation profiles on day of ablation, 28 days from HSCT and once GVHD is diagnosed.
* Patient survival
* Liver function tests
* GVHD grade: skin manifestations, weight, GI and liver histopathology
* Graft-versus-leukemia effect

DETAILED DESCRIPTION:
This study will focus on each individual patient from the early point of myeloablative conditioning through HSCT and GVHD. The rationale for this individualized approach is to account for the anticipated variability in patient age and primary disease, background pathology and individual therapeutic course, considering the enormous heterogeneity of this condition. To compensate for this limitation, we intend to create an individualized algorithm, based on a novel dynamic biomarker, i.e., AAT functionality, individualized per patient and placed on a timeline, with the aim of minimizing future occurrences of GVHD, and by using readily available laboratory measurements. The study is designed around patient sample collection, there is no change in standard of care, therefore there is no intervention as well.

Three types of sample tubes will be collected per indicated time point:

* Serum tube for protein levels and enzymatic activity assays.
* EDTA tube for isolation of peripheral blood mononuclear cells (PBMCs), cells will be stimulated and then analyzed by FACS and lysed for RT-PCR
* EDTA tube for whole blood stimulation assay for further FACS analysis and cytokine production measurement.

After donor and recipient informed consent forms were signed, a single blood sample should be obtained from the donor on the day of transplant extraction. Time points for recipient's samples include the day of myeloablation and again immediately prior to HSCT (set as day 0 and possibly -3 in MUDs). Serum and lysed blood samples will be collected on days 7, 14, 28, and every 21 days thereafter, through the development and progression of GVHD (where relevant). Blood samples for FACS will be collected by days 0 and 28. Sample collection is planned to end within 1 year from HSCT, or two months after appearance of symptoms of GVHD, or two months after a change is introduced in the immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for allogeneic transplantation for the first time, scheduled to receive HSCT from HLA-matched sibling or an unrelated matched donor
* Signed informed consent by the donor(Healthy volunteers) and the patient

Exclusion Criteria:

* Patients undergoing immunosuppressive treatment prior to preparation for bone-marrow transplantation.
* Pregnant and disabled patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In every medical center in which a bone marrow transplantation is performed, allogeneic transplantation recipients will be recruited for the trial.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-01-27 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients progressing into acute or chronic GVHD | Up to 1 year
  Evaluation of patient circulating alpha-1-antitrypsin levels and enzymatic functions as a bio-marker for GVHD progression and grading

SECONDARY OUTCOMES:
Correlation between AAT pattern and survivability, response to immunosuppressive treatment. liver functions, immunocyte activities. | Up to 1 year
  Correlation between AAT patterns and:
  * Circulating immune cell activation profiles on day of ablation, 28 days from HSCT and once GVHD is diagnosed.
  * Patient survival
  * Liver function tests
  * GVHD grade: skin manifestations, weight, GI and liver histopathology
  * Graft-versus-leukemia effect

CONTACTS AND LOCATIONS:
Overall Officials: Eli Lewis, Professor, Principal Investigator — Ben-Gurion University of the Negev
Locations (4):
- Israel (4):
  - Hadassah, Jerusalem, Center
  - Tel Aviv Sourasky Medical Center - Ichilov Hospital, Tel Aviv, Center
  - Rambam MC, Haifa, North
  - Soroka Medical Center, Beersheba, South

IPD SHARING:
Plan to Share IPD: Yes
The clinical individual participant data will be further analyzed by other researchers after the study is completed.That is in order to combine this clinical data with other experiments' results. no